CLINICAL TRIAL: NCT01903538
Title: Interference With Cognitive Control by Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Professor, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 211/2010BO1_2
Record Dates: First submitted 2013-07-13; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cathodal transcranial direct current stimulation (Experimental)
  Interventions: Device: Cathodal transcranial direct current stimulation (tDCS)
- Sham transcranial direct current stimulation (Sham Comparator)
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Cathodal transcranial direct current stimulation (tDCS) — Cathodal transcranial direct current stimulation (tDCS) 20min, 1mA, F3 (EEG 10/20), reference right M. deltoideus
  Arms: Cathodal transcranial direct current stimulation
Device: Sham transcranial direct current stimulation — Sham transcranial direct current stimulation (tDCS) 40s, 1mA, F3 (EEG 10/20), reference right M. deltoideus
  Arms: Sham transcranial direct current stimulation

SUMMARY:
Insufficient cognitive control over emotional distracters is characteristic for major depressive disorder (MDD). Hypoactivation of the dorsolateral prefrontal cortex (dlPFC) is associated with this deficit. In this study the investigators assess the effect of a decrease of dlPFC activity in healthy subjects by cathodal transcranial direct current stimulation (tDCS) on cognitive control.

In a double-blinded, balanced randomized, sham-controlled crossover trial the investigators determine the effect of a single-session of cathodal tDCS to the left dlPFC on cognitive control in healthy subjects. To assess the cognitive control the investigators use a delayed response working memory task (DWM)and an arithmetic inhibition task (AIT) with pictures of varying valence.

ELIGIBILITY:
Inclusion Criteria:

informed consent

Exclusion Criteria:

psychiatric or neurological disorders seizures cardiac pacemakers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Correctness and reaction time of response | Within 30 min starting 5 min after the initiation of stimulation
  Correctness is defined as the percentage of correct responses in the DWM and AIT

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Tübingen, Tübingen, Germany